CLINICAL TRIAL: NCT02362685
Title: Exercise Testing in Metabolic Myopathies
Brief Title: Metabolic Exercise Testing
Acronym: RANNOU
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Principal Investigator, RANNOU, MD, PhD, University Hospital, Brest
Other Study IDs: RANNOU
Record Dates: First submitted 2015-02-04; First posted 2015-02-13 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Metabolic Myopathies; Exercise Test; Myalgia
Keywords: Metabolic myopathies; Exercise testing; Blood sample; Muscle biopsy; Genetic analysis; Cycloergometer; Grip-test; Exercise physiology; Muscle physiology
MeSH Terms: conditions — Myalgia | interventions — Phenotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample Urine sample Muscle tissue DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- metabolic exercise testing: All the subjects referred to performed a metabolic exercise testing.
  Interventions: Device: functional test; Genetic: matching genotype with phenotype

INTERVENTIONS:
Device: functional test — subjects perform a metabolic exercise testing
Genetic: matching genotype with phenotype

SUMMARY:
Exertional symptoms are the hallmarks of metabolic myopathies, supporting the concept of using functional tests when this diagnosis is suspected. Exercise increases the concentration of muscle metabolites in the venous blood supply (e.g. lactate, pyruvate, and ammonia) especially during recovery. The purpose of this study is to compare the results of exercise testing with to the data from muscle biopsy or genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the Physiology Department of Brest Hospital for a metabolic exercise test
* Ability to provide informed consent

Exclusion Criteria:

* Contraindication(s) to perform cardiopulmonary exercise testing (ATS/ACCP statement on cardiopulmonary exercise testing, Am J respi Care Med 167: 211-77, 2003)
* Pregnancy or unknown pregnancy status.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects referred to perform a metabolic exercise testing.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-09; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Whole-body dynamic exercise | Participants will be followed for an expected average of 1 year to determine whether a muscle biopsy is performed
  The relation between Cardiopulmonary exercise test variables and the results of muscle biopsy or genetic analysis will be evaluated.
Grip-test | Participants will be followed for an expected average of 1 year to determine whether a muscle biopsy is performed
  The relation between Grip-test variables and the results of muscle biopsy or genetic analysis will be evaluated.
Blood tests | Participants will be followed for an expected average of 1 year to determine whether a muscle biopsy is performed
  The results of blood analysis from samples performed before, during, and after exercise will be compared to the results of muscle biopsy or genetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Rannou, MD, PhD, Principal Investigator — CHRU Brest
Locations (1):
- Centre Hospitalier Régional Universitaire, Brest, France